CLINICAL TRIAL: NCT05697757
Title: Effects of Dynamic Lighting on Improving Sleep and Mood in Older Adults With Dementia.
Brief Title: Lighting for Older Adults With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Arizona Alzheimer's Consortium (Unknown); Arizona State University Knowledge Enterprise (Unknown)
Responsible Party: Principal Investigator, Nina Sharp, Assistant Professor, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: STUDY00016960
Record Dates: First submitted 2023-01-15; First posted 2023-01-26 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Sleep; Mood
Keywords: Dynamic Lighting; Sleep; Mood; Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Investigators will examine a series of participants (N=30), each of whom will participate in a seven-week experiment. The study will be conducted over seven successive one-week periods with two cohorts of participants experiencing the same series of lighting interventions in a counterbalanced manner.
Who Masked: Participant, Care Provider
Masking Description: Neither participants nor their caregivers will be told about the structure of the lighting conditions and the potential effects, just that the lighting could change daily.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Condition followed by Dynamic Condition (Experimental): Each lighting condition will last for three weeks (Weeks 2-4 or 5-7). The order of conditions will be randomized. Sleep data will be collected only on the last 7 days of each condition using actigraphy. Light spectrum and intensity will be tracked continuously throughout the waking hours (wearable light tracker). Moreover, caregivers will complete two questionnaires (CSDD and CMAI) every seven days to assess the short and long-term effects of each condition on mood and agitation of older adult participants.
  Interventions: Other: Dynamic Lighting; Other: Placebo Lighting
- Dynamic Condition followed by Placebo Condition (Experimental): Each lighting condition will last for three weeks (Weeks 2-4 or 5-7). The order of conditions will be randomized. Sleep data will be collected only on the last 7 days of each condition using actigraphy. Light spectrum and intensity will be tracked continuously throughout the waking hours (wearable light tracker). Moreover, caregivers will complete two questionnaires (CSDD and CMAI) every seven days to assess the short and long-term effects of each condition on mood and agitation of older adult participants.
  Interventions: Other: Dynamic Lighting; Other: Placebo Lighting

INTERVENTIONS:
Other: Dynamic Lighting — This will be an eighteen-hour lighting scheme that includes three modes: morning (6:00 - 12:00), afternoon (12:00 - 18:00), and evening (18:00 - 24:00). It mimics natural lighting by providing blue-enriched high-intensity lighting in the morning and neutral white medium-intensity lighting in the afternoon to maintain alertness without exerting substantial circadian effects. The biodynamic lighting will provide yellowish low-intensity lighting in the evening to minimize any circadian effect.
Other: Placebo Lighting — We will include an active placebo condition that will be a whole-day lighting scheme with constant color and brightness from morning to evening. The numbers of CCT and illuminance levels are selected based on the average room lighting

SUMMARY:
This study aims to investigate the effect of a dynamic lighting intervention on sleep quality, circadian activity rhythms, and mood in older adults with dementia living in long-term care facilities. The dynamic lighting intervention is designed to create an ambient illumination that provides a high level of circadian stimulation in the morning and circadian-neutral lighting in the evenings through delivering varying light intensity and spectrum.

DETAILED DESCRIPTION:
Light is the most important environmental element that is not only necessary to fulfill visual tasks but also is the main stimulus that regulates circadian rhythms. Daily exposure to proper lighting at the right time is reported as an effective non-pharmacological treatment to improve sleep disorders in various age groups including older adults. Several clinical studies have demonstrated the benefits of bright light therapy to improve sleep duration and sleep efficiency at night and reduce daytime sleepiness and behavioral disturbance (i.e., agitation, depression) in older adults. In most of these studies, lighting intervention includes a lightbox that exposes participants to an extra lighting source with specific characteristics (i.e., blue-enriched bright light) for only a few hours without considering the impacts of other lighting sources that individuals are exposed to throughout the day. A significant impediment to administrating bright light therapy for older adults with dementia is that these individuals typically require reminders to remain seated and awake in front of a lightbox long enough to benefit from the bright light exposure. An alternative way to deliver bright light is through providing circadian-effective ambient lighting. The circadian system responds best to high-intensity short-wavelength light (peak wavelength of 480 nm). However, the lighting design in long-term care facilities does not necessarily provide adequate intensity and spectrum to stimulate circadian rhythms in elder residences. Studies reported poor lighting conditions in nursing homes. According to these studies, daytime lighting in these institutions is not even sufficient to fulfill older adults' visual needs, while light at night is relatively often excessive. Thus, this study will be carried out to achieve the following aims:

Aim1: Investigate the effect of a dynamic lighting condition on circadian activity rhythms and selected sleep parameters in older adults with dementia.

Aim2: Evaluate the effect of a dynamic lighting condition on mood.

Findings from this study will provide initial guidance to the designers and administration of memory care facilities as to the lighting design recommendations of greatest benefits to the sleep, mood, and well-being of institutionalized older adults diagnosed with dementia.

The participants will be recruited from two memory care facilities from the greater Phoenix area, based on the recommendation of the managers at the memory care facilities.

Environment: In this study, the human-lighting interaction will occur in the common areas of the selected memory care facilities where older adults with dementia spend most of the daytime hours under the supervision of facility caregivers. Research personnel will install experimental luminaires in the memory care facility's common area. During this visit, research personnel will also give a number of actigraphs and light trackers (which will be used for data collection throughout the study) to caregivers and instruct them on how to use these devices on participants. Participants will also be instructed (by caregivers) on how to use each device.

Week 1 (Baseline): Patterns of sleep, moods, and light exposure will be monitored ad libitum for one week. The experimental luminaires will remain off during Week 1. Placing luminaires in the common area of the facility prior to the use of lighting interventions during Weeks 2 to 7 will minimize environmental variations between baseline and intervention measurements (e.g., new luminaires in the room) and decrease the bias resulting from the Hawthorne effect on collected data.

Weeks 2-7 (Intervention): The intervention period will start right after the baseline and continue for six constructive weeks. There are two lighting interventions, each of which is three weeks long. We will randomly assign one of the residences to start with (Dynamic > Placebo) lighting intervention while the other start with (Placebo > Dynamic) lighting intervention. Actigraphy will be conducted only on the last 7 days of each condition. Light spectrum and intensity will be tracked continuously throughout the waking hours (Blue Iris mobile sensor). Moreover, caregivers will complete CSDD and CMAI every seven days to assess the short and long-term effects of each condition on mood and agitation of older adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 50.
* Diagnosed with mild to major dementia based on the physician and care facility manager's recommendation.
* Has no major organ failure, major diagnosis other than dementia, history of head injury, obstructing cataracts, macular degeneration, and blindness based on their Medical history.
* Not taking light therapy
* Female or male
* No current or planned use of light-altering devices (e.g., blue-blocking and/or tinted glasses and contact lenses)

Inclusion Criteria:

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Nocturnal Sleep Duration (in minutes) as measured by actigraphy | 24 hours everyday during the last 7 days of each condition, namely 7 days of baseline, 7 days of dynamic, and 7 days of placebo.
  Nocturnal Sleep Duration (in minutes) will be measured by Actigraphy. Longer sleep duration corresponds to improved sleep outcomes.
Change in Percent Sleep Efficiency (total sleep time divided by time in bed) measured by actigraphy. | 24 hours everyday during the last 7 days of each condition, namely 7 days of baseline, 7 days of dynamic, and 7 days of placebo.
  Percent Sleep Efficiency will be measured by actigraphy. Higher percentage corresponds to higher sleep quality.
Minutes of wake after sleep onset measured by actigraphy. | 24 hours everyday during the last 7 days of each condition, namely 7 days of baseline, 7 days of dynamic, and 7 days of placebo.
  Minutes of wake after sleep onset will be measured by actigraphy. Lower number indicates better sleep pattern and sleep outcomes.
Changes in depression levels as measured by Cornell Scale of Depression in Dementia (CSDD). | Every seven days throughout the 7-week protocol.
  Depression level is assessed using CSDD every 7 days throughout the 7-week protocol based on caregivers' observations of the participants' behavior during the week prior. Lower scores in CSDD indicates lower depression and better mood outcomes.
Changes in agitation levels measured by Cohen-Mansfield Agitation Inventory (CMAI). | Every seven days throughout the 7-week protocol.
  Agitation level is assessed using CMAI every 7 days throughout the 7-week protocol based on caregivers' observations of the participants' behavior during the week prior. A lower score indicates lower levels of agitations and an improvement in mood.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Sharp, PhD, Principal Investigator — Arizona State University
Locations (3):
- United States (3):
  - Sunshine Village, Phoenix, Arizona
  - ASU DeSmart Lab, Tempe, Arizona
  - Mirabella at ASU, Tempe, Arizona

IPD SHARING:
Plan to Share IPD: Yes
No individual participant data will be shared. Results will be published by the investigators in academic journals and conference proceedings. However, neither the name nor identity of the participants will be used in any publications. Sharing of generated study data will be carried out in several different ways. We plan to make our results available to researchers and potential collaborators interested in human-light interactions.
Time Frame: The data will be available after the data collection and analysis is complete which is anticipated to be in January 2024. The findings will be published in academic journals

REFERENCES:
- [Derived] Alrahyani M, Youngstedt S, Fani M, Yague N, Yu F, Guest MA, Yeom D, Sharp N. Effects of applying biodynamic lighting on improving sleep, depression, and agitation in older adults with dementia: a pilot clinical trial. Geriatr Nurs. 2025 Jul-Aug;64:103435. doi: 10.1016/j.gerinurse.2025.103435. Epub 2025 Jul 4. PMID 40617163